CLINICAL TRIAL: NCT02340156
Title: Phase II Study of Combined Temozolomide and Targeted P53 Gene Therapy (SGT-53) for Treatment of Patients With Recurrent Glioblastoma
Brief Title: Phase II Study of Combined Temozolomide and SGT-53 for Treatment of Recurrent Glioblastoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: SynerGene Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SGT53-02-2
Record Dates: First submitted 2014-12-18; First posted 2015-01-16 (Estimated); Results first posted 2021-03-03 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-02

CONDITIONS: RECURRENT GLIOBLASTOMA
MeSH Terms: conditions — Glioblastoma | interventions — Temozolomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SGT-53 with Temozolomide (Experimental): SGT-53, at 3.6 mg DNA/infusion, will be administered twice weekly in a 28 day cycle starting on Day 1 (cycle 1), Day 29 (cycle 2) and Day 57 (cycle 3). Temozolomide (TMZ) will be administered by mouth daily on days 9-13 of each cycle. Patients who are responding to treatment may receive three additional cycles of SGT-53/TMZ therapy or continue on TMZ alone at investigator's discretion. Surgical resection of recurrent or progressive tumor for tumor analysis is an optional procedure. In these individuals SGT-53, at 3.6 mg DNA/infusion, will be administered twice (on days -1 and -3) in the week prior to surgery. Surgical resection is Day 0. 14-21 days post operatively and having recovered from the effects of surgery, the patients will then start cyclical TMZ with SGT-53 as described above.
  Interventions: Genetic: SGT-53; Drug: Temozolomide

INTERVENTIONS:
Genetic: SGT-53 — SGT-53, at 3.6 mg DNA per infusion, will be administered twice per week for 3 weeks (on Day 1, 4, 8, 11, 15 and 18 of each cycle) for 3 cycles. If SGT-53-related toxicity occurs, the dose of SGT-53 will be de-escalated to 2.4 or 1.2 mg DNA/infusion when appropriate.
Drug: Temozolomide — TMZ will be administered orally on days 9-13 of each cycle. In cycle 1, the dose of TMZ will be 150 mg/m². If the TMZ-related toxicities are tolerated in cycle 1, the dose of TMZ will be escalated to 200 mg/m² for cycle 2 and beyond. If TMZ-related toxicity occurs, the dose if TMZ will be de-escalated to 125 mg/m² (dose level -1), 100 mg/m² (dose level -2) or 75 mg/m² (dose level -3) when appropriate.
  Other Names: Temodar

SUMMARY:
This Phase II clinical trial is an open label, single arm, multicenter study of the combination of intravenously administered SGT-53 and oral temozolomide in patients with confirmed glioblastoma who have proven tumor recurrence or progression. The objective of this trial is to assess 6 month progression free survival (PFS), overall survival (OS), anti-tumor activity, safety and possibly to evaluate, nanoparticle delivery to tumor site, and the induction of apoptosis in the tumor..

DETAILED DESCRIPTION:
The p53 is a vital human tumor suppressor gene. Loss of p53 suppressor function is present in the majority of human cancers. The p53 protein has a diverse range of functions including regulation of cell cycle checkpoints, cell death (apoptosis), senescence, DNA repair, maintenance of genomic integrity, and control of angiogenesis. Abnormalities of the p53 gene may impact the efficacy of standard anticancer treatments such as radiation and chemotherapy. P53 mutation and pathway dysfunction are associated with poor clinical outcomes and the presence of the p53 mutation correlates with resistance to chemotherapy and radiation. The development of somatic gene therapy has created the potential to restore wild type function of p53. SGT-53 is a complex of cationic liposome encapsulating a normal human wild type p53 DNA sequence in a plasmid backbone. This complex has been shown to efficiently and specifically deliver the p53 cDNA to the tumor cells and to cross the blood-brain barrier. Introduction of the p53 cDNA sequence is expected to restore wtp53 function in the apoptotic pathway. P53 restoration has been shown most effective in enhancing cytotoxicity in combination with an agent which results in DNA damage or initiates apoptosis. The primary mechanism of resistance to current standard chemotherapeutic agent Temozolomide (TMZ) is overexpression of O6-methylguanine-DNA-methyl transferase (MGMT), which repairs the TMZ-induced DNA lesion by removing the o6-guanine adducts. Thus, a means to down modulate MGMT activity would enhance the therapeutic effect of TMZ. A number of reports have indicated that increasing wtp53 expression can down-regulate expression of DNA repair genes such as MGMT and increases the sensitivity of tumor cells to alkylating agents. This is a Phase II clinical trial of the tumor-targeted SGT-53 nanocomplex in combination with chemotherapeutic agent, temozolomide which is the standard of care for Glioblastoma Multiforme (GBM) brain tumors. We propose to test the combination of SGT-53 and standard temozolomide to determine efficacy and safety in patients with confirmed glioblastoma who have proven tumor recurrence or progression.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed glioblastoma or gliosarcoma in 1st, 2nd or 3rd relapse.
* Radiographic demonstration of disease progression following prior therapy
* Measurable disease on MRI performed within 14 days prior to registration.
* Male or female patients ≥ 18 years of age.
* Recurrent disease with an:

  * interval of ≥ 3 months following radiotherapy + TMZ;
  * interval of ≥ 14 days between end of surgery and start of protocol therapy for patients who have undergone surgery for recurrent disease.
* Patients who tolerated previous administration with TMZ
* Recovery from the effects of prior therapy:

  * 4 weeks from cytotoxic agents
  * 6 weeks from nitrosoureas
  * 4 weeks from any investigational agent
  * 1 week from non-cytotoxic agents
  * 12 weeks from radiotherapy
* Karnofsky performance status ≥ 60%.
* Complete blood count/differential at screening with adequate bone marrow function
* If patient is receiving steroids, must be on stable or decreasing steroid dose within 5 days prior to treatment initiation with SGT-53.
* Patients must be willing to forego other cytotoxic and non-cytotoxic drug or radiation therapy against the tumor while enrolled in the study.
* Women of childbearing potential must have a negative serum beta-HCG pregnancy test documented within 3 days prior to study initiation.
* Women of childbearing potential must agree to use two reliable methods of contraception from screening and up to 30 days after discontinuation of study treatment
* Males not naturally or surgically sterile, who have a female partner of childbearing potential, must agree to use two reliable methods of contraception from screening and up to 30 days after discontinuation of study treatment
* Acceptable liver function
* Acceptable blood sugar control
* Urinalysis: No clinically significant abnormalities.
* PT and PTT ≤ 1.5 X ULN
* Have recovered from any previous therapy side effects or toxicities
* Organ function characterized by ≤ Grade 1

Exclusion Criteria:

* Histology other than astrocytoma grade IV
* Tumor foci detected below the tentorium or beyond the cranial vault.
* Glioblastoma or gliosarcoma disease with leptomeningeal spread.
* Patients with a history of any other cancer, unless in complete remission, and off all therapy for that disease for a minimum of 5 years
* Patients with serum aspartate aminotransferase, alanine aminotransferase > 2.5 X the upper limit of normal (ULN) and bilirubin >1.5 ULN
* Moderate to severe hepatic impairment.
* Positive results from HIV serology testing, if any available.
* Supine systolic blood pressure < 100 mmHg or supine diastolic blood pressure < 50 mmHg at screening and baseline
* Renal insufficiency or serum creatinine >1.5 X ULN at screening.
* Females who are pregnant or lactating or plan to become pregnant during the course of this study.
* Substance or alcohol abuse or dependence, within 12 months prior to screening.
* Prior chemotherapy for recurrent GBM with nitrosourea compounds including Gliadel® wafers or bevacizumab.
* Prior focal radiotherapy within 3 months of screening.
* Planned treatment, or treatment with any investigational drug within 4 weeks prior to screening.
* Severe, active co-morbidity
* Patients who are currently taking Coumadin or Coumadin derivatives other than to maintain patency of venous access lines.
* Requiring renal dialysis
* Receiving hematopoietic growth factors
* Have significant baseline neuropathies
* Had prior exposure to gene vector delivery products within 6 months
* Any condition that prevents compliance with the protocol or adherence to therapy.
* Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy.
* Treated with antibiotics for infection within one week prior to study entry.
* Fever (> 38.1°C)
* Have diastolic blood pressure of > 90 mm Hg resting at baseline despite medication.
* Serious nonmalignant disease
* Enrollment in a concomitant clinical study
* Have a history of hypersensitivity reaction to any of the components of Temozolomide
* Have a history of hypersensitivity to dacarbazine (DTIC)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-12; Primary Completion 2018-11 (Actual); Study Completion 2018-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John deGroot, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (2):
- MD Anderson Cancer Center, Houston, Texas, United States
- China Medical University Hospital, Taichung, Taiwan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was opened in Houston, Texas, USA and Taichung, Taiwan.
Pre-assignment Details: Only one arm in this study.
Groups:
- SGT-53 With Temozolomide: SGT-53, at 3.6 mg DNA/infusion, will be administered twice weekly in a 28 day cycle starting on Day 1 (cycle 1), Day 29 (cycle 2) and Day 57 (cycle 3). Temozolomide (TMZ) will be administered by mouth daily on days 9-13 of each cycle.
  If SGT-53-related toxicity occurs, the dose of SGT-53 will be de-escalated to 2.4 or 1.2 mg DNA/infusion when appropriate.
  Temozolomide: In cycle 1, the dose of TMZ will be 150 mg/m². If the TMZ-related toxicities are tolerated in cycle 1, the dose of TMZ will be escalated to 200 mg/m² for cycle 2 and beyond. If TMZ-related toxicity occurs, the dose if TMZ will be de-escalated to 125 mg/m² (dose level -1), 100 mg/m² (dose level -2) or 75 mg/m² (dose level -3) when appropriate.
Period: Overall Study
Arm/Group | SGT-53 With Temozolomide
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- SGT-53 With Temozolomide: SGT-53, at 3.6 mg DNA/infusion, will be administered twice weekly in a 28 day cycle starting on Day 1 (cycle 1), Day 29 (cycle 2) and Day 57 (cycle 3). Temozolomide (TMZ) will be administered by mouth daily on days 9-13 of each cycle.
Arm/Group | SGT-53 With Temozolomide
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 60 [60 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Taiwan | 1
Number of Relapse [Count of Participants; unit: Participants]
  First | 1
  Second | 0
  Third | 0

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response
Description: The 6 month progression-free survival (PFS) was evaluated using RANO Response Criteria.
Time Frame: 6 months
Population: The number of participant was too small to analyze.
Groups:
- SGT-53 With Temozolomide: SGT-53, at 3.6 mg DNA/infusion, was administered twice weekly in a 28 day cycle starting on Day 1 (cycle 1), Day 29 (cycle 2) and Day 57 (cycle 3). Temozolomide (TMZ) was administered by mouth daily on days 9-13 of each cycle.
Arm/Group | SGT-53 With Temozolomide
Number analyzed (Participants) | 0

2. Secondary Outcome: Incidence of Treatment-Emergent Adverse Events
Description: The safety of the combination of SGT-53 and Temozolomide was assessed by analysis of adverse experiences, clinical laboratory tests and physical examinations.
Time Frame: Study drug initiation through 30 days after the last dose of study drug or EOS, whichever is later, approximately 90 days.
Population: Adverse events that were grade 3 or above
Measure: Number; unit: Participants
Arm/Group | SGT-53 With Temozolomide
Number analyzed (Participants) | 1
Participants
  Seizure | 1
  Electrocardiogram QT corrected interval prolonged | 1
  Skin ulceration | 1

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Progression-free survival is defined as the time from the date of enrollment to the date of disease progression, or death (any cause) on or prior to the clinical cutoff date, whichever occurs earlier. Subjects who do not have disease progression or have not died will be censored at the date of the last tumor assessment on or prior to the clinical cutoff.
Time Frame: From date of registration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 12 months.
Population: The number of participant was too small to analyze.
Arm/Group | SGT-53 With Temozolomide
Number analyzed (Participants) | 0

4. Secondary Outcome: Overall Survival (OS)
Description: Overall survival is defined as the time from the date of enrollment to the date of death from all causes.
Time Frame: From date of registration until the date of death from any cause, assessed up to 180 months.
Population: The number of participant was too small to analyze.
Arm/Group | SGT-53 With Temozolomide
Number analyzed (Participants) | 0

5. Secondary Outcome: Anti-tumor Activity
Description: The anti-tumor activity of the combination of SGT-53 and Temozolomide was determined based upon the RANO criteria.
Time Frame: as for outcome 3
Population: The number of participant was too small to analyze.
Arm/Group | SGT-53 With Temozolomide
Number analyzed (Participants) | 0

6. Secondary Outcome: Induction of Apoptosis
Description: Flow cytometry or histological examination was used to determine the level of apoptosis induced by SGT-53 in tumors resected 3 days after the first SGT-53 infusion (optional procedure)
Time Frame: 3 days
Population: The number of participant was too small to analyze.
Arm/Group | SGT-53 With Temozolomide
Number analyzed (Participants) | 0

7. Secondary Outcome: Nanoparticle Tumor Delivery
Description: As an indicator of nanoparticle delivery to the tumors, DNA PCR was used to determine the presence of SGT-53 delivered exogenous wt p53 in the tumors. This analysis will be performed on any tumors resected 3 days after the first SGT-53 infusion (optional procedure)
Time Frame: 3 days
Population: The number of participant was too small to analyze.
Arm/Group | SGT-53 With Temozolomide
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Study drug initiation through 30 days after the last dose of study drug or End of Study, whichever is later, approximately 90 days.
Arm/Group | SGT-53 With Temozolomide
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SGT-53 With Temozolomide (N=1)
Seizure (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SGT-53 With Temozolomide (N=1)
Electrocardiogram QT corrected interval prolonged (Investigations) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
The number of participant was too small for statistical analysis. The study was terminated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-05): https://cdn.clinicaltrials.gov/large-docs/56/NCT02340156/Prot_SAP_000.pdf